CLINICAL TRIAL: NCT06909760
Title: A Myth Orthopaedic Implant Pain in Cold Weather
Status: Active, not recruiting | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Ahmet Berkay Girgin, Supervisor İnvestigator, Ankara Etlik City Hospital
Other Study IDs: Implant Pain in Cold
Record Dates: First submitted 2025-03-17; First posted 2025-04-03 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-03

CONDITIONS: Pain; Cold Temperature
Keywords: pain; implant; cold weather
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients with orthopaedic implants: The contact information of the patients who volunteered to participate in the study will be obtained and the patients will be called for 2 separate controls based on the one-week average value of the air temperature (2 periods with a one-week average air temperature between 27-35°C (hot weather) and 0-8°C (cold weather)).
  Parameters to be investigated in patients called for control in both weather conditions;
  * Whether there are any complaints at the implant site
  * Visual pain score (VAS)
  * Proximal and distal range of motion (ROM) of the operated extremity
  * Chills/shivering according to the opposite extremity
  * Pain catastrophizing scale (PCS)
  * Measures taken in cold weather
  * The temperature difference between the implant site and the same site in the opposite extremity will be measured using thermal thermometers.

SUMMARY:
In daily practice, the investigators frequently hear patients with orthopaedic implants complaining of implant pain and coldness in the implant area in cold weather in outpatient clinics. However, when the literature is examined, there is only one study examining the effect of cold weather on the implant and only the pain in cold weather was questioned in this study. In this study, the investigators aimed to obtain clearer information by comparing the effect of cold air on orthopaedic implants with hot air with many parameters.

DETAILED DESCRIPTION:
Fractures and degenerative joint diseases are common medical problems that many people experience throughout their lives. Orthopaedic implants are widely manufactured and used worldwide to replace a degenerated joint or to reduce a fractured bone and promote healing (1). In a 1988 incidence study, it was estimated that 4.9 million people in the USA had fixation material (2). Today, this rate is thought to increase much more due to increasing population, developing and increasing number of motorised vehicles and increasing surgical indications. Although the removal of these implants is a very controversial issue in the literature, most surgeons do not recommend routine removal of implants unless there are complications (3). In a study, it was reported that the reasons for implant removal were osteomyelitis and persistent pain in only 28% of patients, but the reason for removal was 'patient request' in 72% of patients who had implants removed (4).

In daily practice, the investigators frequently hear patients with orthopaedic implants complaining of implant pain and coldness in the implant area in cold weather in outpatient clinics. However, when the literature was examined, there was only one study examining the effect of cold weather on the implant and only the pain in cold weather was questioned in this study. In this study, the investigators aimed to obtain clearer information by comparing the effect of cold air on orthopaedic implants with hot air with many parameters.

ELIGIBILITY:
Inclusion Criteria:

* patients aged ≥ 18 years with orthopaedic implants due to orthopaedic trauma.

Exclusion Criteria:

* Patients <18 years of age
* Patients with incomplete fracture union
* Patients with joint prosthesis (knee, hip, shoulder prosthesis, etc.)
* Patients with complications in the operated extremity (implant infection, implant failure, etc.)
* Acute or chronic infection (bacterial or viral infection) of any body site
* Patients diagnosed with neuropathy (diabetic, alcoholism, autoimmune, nutritional deficiency, infectious)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All population
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-05-25 (Estimated)

PRIMARY OUTCOMES:
Pain on the extremity which was operated | Patients are called for follow up twice a year with 6 months interval
  Pain will be assessed with "Visual Analogue Scale". Patients will be asked if they have pain on their extremity with orthopedic implant both in cold and hot weather conditions.

SECONDARY OUTCOMES:
range of motion of the affected joints | Patients are called for follow up twice a year with 6 months interval
  Range of motion of the affected extremities will be evaluated with goniometer. Affected joints mean the joints which is proximal and distal to orthopedic implant used. If there is an implant in tibia. Range of motion of the knee and ankle joints will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmet Acar, Ankara, Turkey (Türkiye)